CLINICAL TRIAL: NCT00147901
Title: Multicenter Phase II Trial of Fludarabine and Cyclophosphamide in Combination With Alemtuzumab (FC-Cam) for Patients With Relapsed Chronic Lymphocytic Leukemia - CLL-2L Protocol of the German CLL-Study Group (GCLLSG)
Brief Title: Fludarabine, Cyclophosphamide, and Alemtuzumab in Patients With B-cell Chronic Lymphatic Leukemia (B-CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: University of Cologne (Other); MedacSchering Onkologie (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL-2L; 2005-003017-32 (EudraCT Number)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: B-cell Chronic Lymphocytic Leukemia
Keywords: CLL; Immunochemotherapy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Cyclophosphamide; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FCCam (Experimental): After an initial subcutaneous dose escalation of alemtuzumab over 2 days, 30 mg alemtuzumab s.c., cyclophosphamide 200 mg/m2 i.v. and 25 mg/m2 fludarabine i.v. were administered on three consecutive days. Treatment was repeated after 28 days for up to six cycles
  Interventions: Drug: FCCam

INTERVENTIONS:
Drug: FCCam — After an initial subcutaneous dose escalation of alemtuzumab over 2 days, 30 mg alemtuzumab s.c., cyclophosphamide 200 mg/m2 i.v. and 25 mg/m2 fludarabine i.v. were administered on three consecutive days. Treatment was repeated after 28 days for up to six cycles
  Other Names: Fludarabine, Cyclophosphamide, Alemtuzumab

SUMMARY:
This study aims to assess the short term efficacy of a combination immunochemotherapy in patients with relapsed B-cell chronic lymphatic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* B-CLL in need of treatment
* One or two prior prior therapies
* WHO performance status 0-2

Exclusion Criteria:

* Serum creatinine > 1.5 ULN
* Major organ dysfunctions
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-01; Primary Completion 2008-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete and partial response rate) | 28 days after the end of the last cycle
  Response Evaluation has to be done according the the NCI guidelines

SECONDARY OUTCOMES:
Toxicity | 28 days following the last dose of FCCam
MRD response rate | 28 days after the end of the last cycle
Response rate in biological defined risk groups | 28 days after the end of the last cycle
Duration of response | up to 36 months after the end of treatment
Treatment administration (dose intensity) | up to the last day of the last given cycle (day 28 of the 6th cycle)
Overall survival | up to 36 months after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elter T, James R, Busch R, Winkler D, Ritgen M, Bottcher S, Kahl C, Gassmann W, Stauch M, Hasan I, Staib P, Fischer K, Fink AM, Bahlo J, Buhler A, Dohner H, Wendtner CM, Stilgenbauer S, Engert A, Hallek M. Fludarabine and cyclophosphamide in combination with alemtuzumab in patients with primary high-risk, relapsed or refractory chronic lymphocytic leukemia. Leukemia. 2012 Dec;26(12):2549-52. doi: 10.1038/leu.2012.129. Epub 2012 May 15. No abstract available. PMID 22584787